CLINICAL TRIAL: NCT04432350
Title: Assessment of Mortality Rates in SARS-CoV-2 Infected Populations Treated With Repurposed Medications
Brief Title: Assessment of Mortality Rates in COVID-19 Infected Populations Treated With Repurposed Medications
Status: Withdrawn | Type: Observational
Why Stopped: Limitations with data.
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID-19_TRHCPrescribeWellness
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: COVID; Drug Effect; Drug Interaction; Risk Reduction
Keywords: COVID-19; Adverse Drug Event; Mortality Rate
MeSH Terms: conditions — Risk Reduction Behavior; COVID-19; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated with Repurposed Drugs: This cohort will be for individuals who have tested positive for COVID-19 and were treated with repurposed drugs. This will be tracked via drug claims data in a PrescribeWellness Pharmacy.
- Not Treated with Repurposed Drugs: This cohort will be for individuals who have tested positive for COVID-19 and were not treated with repurposed drugs. This will be tracked via drug claims data in a PrescribeWellness Pharmacy.

SUMMARY:
This retrospective cohort study will include eligible patients that received a positive COVID-19 test and filled a new prescription for one of the repurposed medications (including hydroxychloroquine, chloroquine, with or without azithromycin) for the treatment of COVID-19 at a PrescribeWellness pharmacy. The study will use de-identified data collected from February 1, 2020 to start of study. The data set will include: repurposed medication name, strength, and dose; age (age limit set at 89 years old); gender; provider type; zip code (excludes 17 three-digit zip code tabulation areas that have a population of 20,000 or fewer persons); conditions; mortality; and a list of concomitant prescriptions.

DETAILED DESCRIPTION:
There is a deficit in literature assessing the risk associated with these repurposed medications in COVID-19 patients. The investigators propose to evaluate if the use of repurposed drugs including hydroxychloroquine and chloroquine is associated with an increased risk of mortality in COVID-19 infected patients treated with such medications.

PrescribeWellness, a Tabula Rasa HealthCare solution, a leading patient relationship management service provider in U.S., facilitates collaboration between more than 15,000 pharmacies and payers, providers, and patients for better health. PrescribeWellness empowers community pharmacies with innovative technological solutions that advance a pharmacist's ability to identify, manage, and drive patient care interventions. On average, 2,000 patients receive their services per each pharmacy. PrescribeWellness expands the medication risk mitigation program of Tabula Rasa HealthCare in community pharmacies and ambulatory patients. The investigators propose to perform a retrospective analysis of data from infected COVID-19 patients served by PrescribeWellness pharmacies for assessing mortality and risk/benefit associated with the use of repurposed COVID-19 drugs.

An approach to reduce and predict adverse drug events is the use of predictive risk scores. Tabula Rasa HealthCare's proprietary MedWise Risk Score™ (MRS) is based on five aggregated medication risk mitigation factors: FAERS (FDA adverse events reporting system) risk score, anticholinergic burden, sedative burden, drug-induced long QT syndrome, and CYP450 drug interaction burden. The MRS™ is a predictive tool used by health care providers to determine which factors, including prescription drugs, can contribute the most to a patient's likelihood of an adverse drug event (ADE) occurring. In order to calculate the MRS™, patient data is first de-identified, and then comprised by various physiological, pharmacological and biochemical variables. Once a patient is analyzed, his/her MRS™ is defined as Very Low, Low, Moderate, High, or Very High Risk for the likelihood of ADE. The investigators propose to retrospectively calculate the MRSTM and assess the predictive value of MRS™ in patients tested positive for COVID-19 and who were treated with repurposed drugs. The investigators hypothesize that an increase rate of mortality is associated with high risk MRS in patients receiving repurposed drugs against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving services at a PrescribeWellness pharmacy;
* Patients who received a COVID-19 positive test at a PrescribeWellness Pharmacy or other certified COVID-19 test centers since February 1, 2020;

Exclusion Criteria:

* Patients who received a COVID-19 negative test at a PrescribeWellness Pharmacy or other certified COVID-19 test centers since February 1, 2020;
* Patients who received COVID-19 repurposed drugs without laboratory-confirmed test for COVID-19 disease;
* Patients who were receiving COVID-19 repurposed drugs prior to February 1, 2020.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PrescribeWellness is a national pharmacy network that serves over 15,000 pharmacies, with an average of over 2,000 patients per pharmacy (~30 million patients). Data will be provided by Tabula Rasa HealthCare PrescribeWellness Analytics department to Tabula Rasa HealthCare's Precision Pharmacotherapy Research & Development Institute. All protected health information (PHI) will be removed from the data set before its transfer through an encrypted server.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
The rate of mortality in patients with a confirmed (positive test result) COVID-19 infection observed by PrescribeWellness pharmacies will be determined. | Six months
  Quantitative
The relationship between high-risk cardio-pulmonary and vascular comorbidities (e.g., hypertension, dyslipidemia, diabetes, and chronic lung diseases) and mortality with use of repurposed medications for the treatment of COVID-19 will be investigated. | Six months
  Quantitative
The MRS™ will be calculated using drug claim data from confirmed COVID-19 patients and explore the predictive value of MRS™ for ADE, LQTS and all-cause of death. | Six months
  Quantitative

SECONDARY OUTCOMES:
To compare the rates of death in COVID-19 confirmed patients treated with repurposed medications versus COVID-19 confirmed patients not treated with repurposed drugs. | 1 year
  Quantitative
The relationship between medications used to treat these underlying health conditions (e.g. ACE inhibitors, angiotensin type 1 receptor blockers, aliskiren, and mineralocorticoid antagonists) and mortality in patients with a confirmed COVID-19 infection. | 1 year
  Quantitative
To compare the MRS™ and its predictive value for ADE between confirmed COVID-19 patients treated with repurposed drugs and confirmed patients not treated with repurposed drugs. | 1 year
  Quantitative
To examine drug regimen patterns associated with higher risk of MRS™, ADEs, and higher rates of death in confirmed COVID-19 patients with and without repurposed medication. | 1 year
  Quantitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu L, Wang B, Yuan T, Chen X, Ao Y, Fitzpatrick T, Li P, Zhou Y, Lin YF, Duan Q, Luo G, Fan S, Lu Y, Feng A, Zhan Y, Liang B, Cai W, Zhang L, Du X, Li L, Shu Y, Zou H. Clinical characteristics of coronavirus disease 2019 (COVID-19) in China: A systematic review and meta-analysis. J Infect. 2020 Jun;80(6):656-665. doi: 10.1016/j.jinf.2020.03.041. Epub 2020 Apr 10. PMID 32283155
- See also: COVID-19 Dashboard — http://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: Coronavirus Dashboard Johns Hopkins — http://coronavirus.jhu.edu/map.html